CLINICAL TRIAL: NCT03595189
Title: Dose Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of an Infusion of Cilastatin in Healthy Volunteers.
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of an Infusion of Cilastatin in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spherium Biomed (Industry)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: SP15016-09; 2017-004795-63 (EudraCT Number)
Record Dates: First submitted 2018-06-18; First posted 2018-07-23 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Dose Finding Study
MeSH Terms: interventions — Cilastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cilastatin Dose 1 (Experimental): Starting dose (3g of Cilastatin) Single intravenous administration during 3 hours.
  Interventions: Drug: Cilastatin
- Cilastatin Dose 2 (Experimental): Dose escalation Single intravenous administration during 3 hours.
  Interventions: Drug: Cilastatin
- Cilastatin Dose 3 (Experimental): Dose escalation Single intravenous administration during 3 hours.
  Interventions: Drug: Cilastatin
- Placebo (Placebo Comparator): Saline solution for infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilastatin — Dose escalation 3-hour single intravenous administration
  Other Names: Cilastatin sodium
  Arms: Cilastatin Dose 1; Cilastatin Dose 2; Cilastatin Dose 3
Drug: Placebo — 3-hour single intravenous administration
  Arms: Placebo

SUMMARY:
This is a phase I, randomized, single-blind, parallel group, placebo-controlled, multi-cohort, first-in-human dose escalation study of a single IV 3-hour administration of Cilastatin as stand-alone in healthy male and female volunteers.

The study objectives are:

The evaluation of safety and tolerability of single intravenous doses of cilastatin in healthy volunteers administered as a 3-hour infusion.

The evaluation of the pharmacokinetic characteristics of Cilastatin after a single 3-hour infusion dose.

DETAILED DESCRIPTION:
The study is designed as a phase I, randomized, single-blind, parallel group, placebo-controlled, multi-cohort, first-in-human dose escalation study of a single IV 3-hour administration of Cilastatin as stand-alone in healthy male and female volunteers.

The study will involve 24 healthy male and female healthy subjects, divided in three study cohorts (8 subjects per cohort). The study is a dose escalating study, starting from 3 g of Cilastatin administered intravenously in 3 hours.

Eight subjects will be randomized and assigned to either the study drug or placebo group for each study cohort in a 3:1 ratio (6 actives and 2 placebos). Randomization will also be gender balanced within each study cohort. The planned dose escalation scheme should not occur before participants in the previous dose level have been treated and safety profile of Cilastatin from those participants are assessed in accordande with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, 18-45 years (inclusive) of age at the time of enrolment.
* Male and female subjects willing and able to give their written consent to participate in the trial after having received information about the study design, the objectives of the project, the possible derivative risks, and their right to withdraw from the study at any time and for any reason.
* Body weight within normal range (Quetelet's index between 19 and 30 expressed as kg/m2 and weigh at least 50 kg and no more than 100 kg inclusive).
* Normal clinical records and physical examination.
* Laboratory tests (hematology, biochemistry and urine analysis) within the range of normal values, per the Biochemistry laboratory reference values of the 'Hospital Universitario La Paz'. Variations may be admitted per the clinical criteria of the clinical investigator.
* Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* To be able to understand the nature of the study and comply with all their requirements.

Exclusion Criteria:

* Women of childbearing potential who planned to become pregnant, were pregnant and/or breast-feeding, or did not wish to use an effective contraceptive method (hormonal contraceptives [implant, patches, oral]) or double-barrier methods [any double combination of: IUD, male or female prophylactics with spermicidal gel, diaphragm, contraceptive sponge, cervical cap]).
* History of alcohol dependence or drug abuse in the last 1 year or daily consumption of alcohol > 40 g/day for men or 24 g/day for women.
* Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day).
* Background of allergy, idiosyncrasy or hypersensitivity to drugs.
* Intake of any medication within 4 days prior and during visit 2 or Xanthine containing foods or beverages or herbal remedies that could interfere with pharmacokinetics of the study drug, except allowed contraceptive medication for female subjects.
* Positive serology for hepatitis B, C or HIV.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, haematological or neurological disease or other chronic diseases.
* Twelve lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
* Having undergone major surgery during the previous 6 months.
* Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc.) from 6 months prior to drug administration.
* Participation in another clinical trial during the 3 months preceding the drug administration.
* Donation of blood during the 4 weeks preceding the drug administration.
* Acute illness within four weeks before drug administration.
* Clinically significant abnormal laboratory values (as determined by the PI) at the screening evaluation.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract
* Positive results of the drugs at screening period or at visit 2. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Benzodiazepines and Cannabinoids (positive results may be repeated at the discretion of the investigator team).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From baseline up to follow-up (approximately 7 days after treatment administration).
Safety measures: Changes in Heart rate values will be assessed for each dose level of cilastatin | From baseline up to follow-up (approximately 7 days after treatment administration).
Safety measures: Changes in Blood pressure values will be assessed for each dose level of cilastatin | From baseline up to follow-up (approximately 7 days after treatment administration).
Safety measures: Changes in Body temperature values will be assessed for each dose level of cilastatin | From baseline up to follow-up (approximately 7 days after treatment administration).
Safety measures: Changes in clinical Laboratory testing will be assessed for each dose level of cilastatin. | From baseline up to follow-up (approximately 7 days after treatment administration)
Safety measures: Changes in Electrocardiogram (ECG) parameters will be assessed for each dose level of cilastatin. | From baseline up to follow-up (approximately 7 days after treatment administration).
  Changes in QTc Interval will be assessed.
Safety measures: Continuous cardiac monitoring (by a holter monitor) will be assessed for each dose level of cilastatin. | From baseline up to 24 h Post-dose
  Changes in electrocardiography heart activity will be assessed.
Assessment of any infusion site reaction | From baseline up to follow-up (approximately 7 days after treatment administration).

SECONDARY OUTCOMES:
Determination of the Area under the curve versus time | From baseline up to 24 hours post start of drug administration
Determination of plasma concentrations | From baseline up to 24 hours post start of drug administration
Determination of renal clearance | From baseline up to 24 hours post start of drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Frías, MD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Clinical Trials Unit, School of Medicine, Universidad Autónoma de Madrid, Madrid, Spain

REFERENCES:
- [Derived] Faubel S. Acute Cardiac Injury Mediates a Distinct Form of CKD: Is This Cardiorenal Syndrome Type 7? J Am Soc Nephrol. 2025 Dec 1;36(12):2317-2319. doi: 10.1681/ASN.0000000905. Epub 2025 Oct 27. No abstract available. PMID 41143893
- [Derived] Funahashi Y, Hebert JF, Munhall A, Aomura D, Burfeind KG, Nguyen ED, Groat T, Nickerson MN, Eiwaz MB, Nelson JW, Andeen NK, Yanagita M, Gurley SB, Hutchens MP. Cardiac LIM Protein, Kidney Fibrosis, and Vascular Change after Acute Cardiorenal Syndrome. J Am Soc Nephrol. 2025 Dec 1;36(12):2330-2347. doi: 10.1681/ASN.0000000774. Epub 2025 Jun 19. PMID 40536823